CLINICAL TRIAL: NCT04146454
Title: A New Smartphone-based Wearable Telerehabilitation System for People With Parkinson's Disease
Brief Title: Smartphone-based Wearable Telerehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Houston (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 16191-01; 1R21HD099242 (NIH)
Record Dates: First submitted 2019-10-16; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; In-home balance training; Smartphone-based wearable telerehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Study participants will be assigned to either of two groups (intervention group and control group)
Who Masked: Investigator
Masking Description: Potential participants diagnosed with Parkinson's disease will be randomly assigned to either of two groups (intervention group and control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone-based balance exercises (Experimental): This group will complete in-home dynamic weight-shifting balance exercises (i.e., physical therapists' recommended dynamic balance exercises) with a smartphone-based wearable telerehabilitation system.
  Interventions: Other: Smartphone-based balance exercises
- Paper-based balance exercises (No Intervention): This group will complete in-home dynamic weight-shifting balance exercises (i.e., physical therapists' recommended dynamic balance exercises) with typical paper-based instructions.

INTERVENTIONS:
Other: Smartphone-based balance exercises — A smartphone-based wearable telerehabilitation system will provide video and audio instructions on how to perform in-home dynamic weight-shifting balance exercises (i.e., physical therapists' recommended dynamic balance exercises).
  Arms: Smartphone-based balance exercises

SUMMARY:
Parkinson's disease (PD), one of the most common neurological disorders, affects at least 10 million people worldwide. The cardinal motor impairments are tremor, bradykinesia, muscle rigidity, and postural instability. While dopaminergic medication and surgical treatment have been shown to suppress tremor, bradykinesia, and muscle rigidity, they do not prevent the progression of the disease or effectively treat postural instability. The latter impairment, which often leads to frequent falls, substantially restricts motor performance and daily activities.

PD is commonly managed in outpatient neurology or movement disorder clinics. Clinical studies have shown that physical and balance rehabilitation regimens supervised by physical therapists can improve postural stability in people with PD for short (hours to days) and long (weeks to months) periods. Cost, limited availability of physical therapists, etc., however, often prohibit many people with PD from undertaking such regimens. Evidence is mounting that periodic and continuous exercising is important for people with PD who are under care at home. Nevertheless, when given a rehabilitation regimen to practice at home, compliance (i.e., adherence) and engagement generally decrease in the absence of real-time therapeutic feedback. The PI has developed a smartphone-based, wearable balance rehabilitation system, known as the Smarter Balance System (SBS), which supplies real-time feedback to people with PD practicing balance rehabilitation regimens at home.

The objectives of this study are to assess and compare the results of long-term rehabilitative balance training for people with PD performing in-home balance training regimens with assistive guidance via the SBS (intervention group) to people following a typical paper-based regimen (control group). The carry-over effects of long-term rehabilitative training by the intervention group and the control group on static/dynamic balance performance, daily activities, and confidence in less fear of falling are analyzed quantitatively and qualitatively.

DETAILED DESCRIPTION:
This study examines static/dynamic balance performance, daily activities, and confidence in less fear of falling for people with Parkinson's disease (PD) performing in-home balance exercises with a smartphone-based wearable telerehabilitation system (intervention group) compared to typical paper-based balance exercises (control group). Twenty-two subjects with idiopathic PD will be randomly assigned to either of two groups of eleven (intervention group (IG) and control group (CG)). The experimental design will include laboratory assessments (i.e., pre-assessment baseline at the beginning of week 1, post-assessment at the end of week 6, and retention-assessment 1 month after week 6) and in-home balance exercises. IG and CG will perform in-home balance exercises (3 days per week for 6 consecutive weeks) with the Smarter Balance System (SBS) recently developed by the PI or the paper-based regimen, respectively. Both groups will also use Fitbits for 6 weeks.

Laboratory assessments: Subjects will be quantitatively assessed for static/dynamic balance performance using a measure for the range of limits of stability (LOS) in both anterior-posterior (A/P) and medial-lateral (M/L) directions, and a Sensory Organization Test (SOT) consisting of six conditions (1: Normal vision and fixed support; 2: Absent vision and fixed support; 3: Sway-referenced vision and fixed support; 4: Normal vision and sway-referenced support; 5: Sway-referenced support and absent vision; and 6: Sway-referenced vision and sway-referenced support) using a Balance Master® (NeuroCom International Inc., USA). During the SOT, center of pressure (COP) data as a function of the six SOT conditions will be collected at a rate of 100 Hz for postural sway analysis. After the completion of quantitative balance assessments, balance performance will be qualitatively assessed using the Activities-specific Balance Confidence (ABC) scale and the Falls Efficacy Scale (FES). A modified Community Health Activities Model Program for Seniors (CHAMPS) will be used to collect the levels of exercise and non-exercise physical activity. After completion of the pre-assessment, a member of the research team will train subjects to use the SBS's smartphone and the Fitbit. Only the IG will be additionally trained in the use of the custom belt and the walker and multimodal biofeedback for in-home dynamic WSBE guided by the SBS. For CG subjects, the physical therapist (Co-I) will review the paper-based regimen for in-home dynamic WSBE. After completion of the post-assessment, only the IG will complete a usability and acceptability questionnaire (UAQ) for the SBS.

In-home balance exercises: Both groups will use the SBSs and Fitbits for 6 consecutive weeks. Only the IG will complete in-home dynamic weight-shifting balance exercises (i.e., physical therapists' recommended dynamic balance exercises, hereafter dynamic WSBE) with the SBS (3 days per week). The CG will perform dynamic WSBE following the paper-based regimen (3 days per week) in accordance with the Health Professionals' Guide to the Physical Management of Parkinson's disease, including detailed descriptions regarding stance condition, movements in both A/P and M/L directions, and repetitions. Only the CG will use the SBS's smartphones and the Fitbits (the SBS's custom belt will not be provided to the IG). To assure a safe exercise environment, both groups will perform in-home dynamic WSBE by standing inside a walker (no wheels). For the IG, the instructional video provided by the SBS will show how to perform dynamic WSBE in both A/P and M/L directions by standing inside the walker without touching or holding onto it unless the subject experiences loss of balance. For the CG, paper-based instructions will be provided. Both groups will be instructed to continue taking prescribed PD medication. After each trial, the IG smartphone app will store exercise-related data. The IG and CG smartphones will store physical activity data (daily number of taken steps and associated distance) collected from the Fitbit.

Performance metrics: Measured data from the Balance Master®, the SBSs, and the Fitbits will be analyzed using MATLAB (The MathWorks, USA). As a function of the pre/post/retention-assessments, two primary outcome measures (range of LOS and SOT score) will be used to evaluate static/dynamic balance performance. Ranges of LOS in degrees correspond to the furthest deviations of the body tilt in both A/P and M/L directions. The SOT score that can be directly obtained from the Balance Master® ranges from 0 to 100, where 100 indicates no postural sway and 0 indicates a fall. The four supplementary outcome measures, which are standard metrics for assessing balance performance, are a root mean square of postural sway (RMS sway) in both A/P and M/L directions, elliptical area of postural sway (sway area), and approximate entropy of postural sway (sway ApEn). Both RMS sway and sway area are linear measures of balance performance, and the sway ApEn is a non-linear measure quantifying the complexity and regularity of postural stability. For the IG, the UAQ score (Likert scale) will be used to assess the usability and acceptability of the SBS, and the IG's compliance with the in-home balance training regimens, total exercise time, and number of completed exercises will be quantitatively analyzed. For both groups, daily number of taken steps and associated distance obtained from Fitbits and ABC scale, FES, and CHAMPS score will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50 and 75 years.
2. Diagnosis of idiopathic PD with a score of 2 and 4 on the Hoehn and Yahr scale.
3. Live with family members or have caregivers.
4. Able to provide informed consent.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Cognitive score less than 26 as determined by the Montreal Cognitive Assessment.
3. Are not ready for physical activity as determined by the modified Physical Activity Readiness Questionnaire.
4. Have dyskinesia.
5. Unable to stand independently for 10 minutes due to dyskinesia.
6. Have severe distal sensory loss.
7. Are medically unstable (chest pain upon exertion, dyspnea, or epilepsy).
8. Have any peripheral, neurological, or musculoskeletal conditions other than PD.

   1. History of peripheral sensory disease that might affect balance stability (e.g., peripheral neuropathy, Type 2 diabetes, vestibular disorder, etc.).
   2. History of central neurologic dysfunction such as stroke or myelopathy.
   3. History of functionally significant musculoskeletal dysfunction (e.g., lower extremity total joint replacement in the past six months, lower extremity fracture/sprain in the past six months, limited ankle range of motion (ankle dorsiflexor/plantar flexor weakness or great toe weakness), etc.).
9. Body mass index (BMI) over 35 computed from individual's height and weight.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Range of limits of stability; change is being assessed | Pre-assessment (baseline at the beginning of week 1)
  Limit of stability refers to the outermost range in anterior-posterior and medial-lateral directions at which the subject can lean from the vertical without changing the base of support. A higher range of limits of stability indicates better balance performance.
Sensory Organization Test (SOT) score; change is being assessed | Pre-assessment (baseline at the beginning of week 1)
  Sensory Organization Test (SOT) score ranges from 0 to 100, where 100 indicates no postural sway and 0 indicates a fall.
Root mean square (RMS) of postural sway; change is being assessed | Pre-assessment (baseline at the beginning of week 1)
  Root mean square (RMS) of postural sway is the primary measure of postural sway. A lower value of root mean square (RMS) of postural sway indicates more stable balance.
Elliptical area of postural sway; change is being assessed | Pre-assessment (baseline at the beginning of week 1)
  Elliptical area of postural sway is the area of postural sway. Smaller sway area indicates better balance performance.
Approximate entropy of postural sway; change is being assessed | Pre-assessment (baseline at the beginning of week 1)
  Approximate entropy of postural sway refers to the complexity and regularity of postural sway. It ranges from 0 to 2, where 0 indicates regular postural sway and 2 indicates complexity postural sway.

SECONDARY OUTCOMES:
Activities-specific Balance Confidence (ABC) scale | Pre-assessment (baseline at the beginning of week 1), post-assessment (at the end of week 6), and retention-assessment (1 month after week 6)
  The Activities-specific Balance Confidence (ABC) scale is a 16-item self-reported measure used by subjects to rate their balance confidence in performing activities. The minimum and maximum scores are 0 and 100; a score of zero represents no confidence in balance, and a score of 100 represents complete confidence in balance.
Fall Efficacy Scale (FES) | Pre-assessment (baseline at the beginning of week 1), post-assessment (at the end of week 6), and retention-assessment (1 month after week 6)
  The Fall Efficacy Scale (FES) is a self-reported questionnaire consisting of a 10 item rating scale used by subjects to rate their balance confidence in performing daily activities without falling. The Fall Efficacy Scale (FES) has a scale from 1 to 10, with 1 being very confident in performing daily activities without falling and 10 being not confident at all in performing daily activities without falling.
Community Health Activities Model Program for Seniors (CHAMPS) | Pre-assessment (baseline at the beginning of week 1), post-assessment (at the end of week 6), and retention-assessment (1 month after week 6)
  The Community Health Activities Model Program for Seniors (CHAMPS) is a self-reported physical activity questionnaire. The minimum and maximum scores are 0 and 41; a higher score indicates better physical activity.

OTHER OUTCOMES:
Usability and acceptability questionnaire (UAQ) | Post-assessment (at the end of week 6)
  The Usability and acceptability questionnaire (UAQ) is a self-reported questionnaire used by subjects to assess the usability and acceptability of the proposed smartphone-based wearable telerehabilitation system. The Usability and acceptability questionnaire (UAQ) has a scale from 24 to 120, with 120 being very confident in using the system and 24 being not confident at all in using the system.

CONTACTS AND LOCATIONS:
Overall Officials: Beom Chan Lee, PhD, Principal Investigator — University of Houston
Locations (1):
- Center for Neuromotor and Biomechanics Research, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All of the materials collected are for research purposes only, and all data will be kept in strict confidence. No information will be given to anyone without permission from the subject. The consent form includes the informed consent statement required by University of Houston IRB for studies involving human subjects. This statement guarantees confidentiality and identifies the subject as the owner of information we collected from this study. Confidentiality will be ensured by use of identification codes. All data, whether generated in the laboratory or at the subject's home, will be identified with an identification code unique to the subject.